CLINICAL TRIAL: NCT01697904
Title: Randomized Trial of a Limited Versus Traditional Oxygen Strategy During Resuscitation in Premature Newborns
Brief Title: Trial of a Limited Versus Traditional Oxygen Strategy During Resuscitation in Premature Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Vishal Kapadia, Assistant Professor of Pediatrics, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 052011-044
Record Dates: First submitted 2012-09-25; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Prematurity; Oxidative Stress
MeSH Terms: conditions — Premature Birth | interventions — Delivery Rooms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Oxygen Strategy (Experimental): Resuscitation was initiated with room air (21% O2) for LOX infants. Supplemental oxygen was given if 1) the heart rate (HR) was less than 100 bpm after 30 seconds of effective ventilation, 2) the lower limits of goal saturations were not met. Targeted goal Pre-ductal saturations after birth were derived by approximation of the interquartile values for healthy term infants as reported by Kamlin et al and Dawson et al.FiO2 was increased or decreased by 10% in 30 second intervals as needed. If HR < 60 bpm after 30 seconds of effective ventilation , FiO2 was increased to 100% until the heart rate was stabilized.
  Targeted Pre-ductal SpO2 After birth
  1. min 60%-65%
  2. min 65%-70%
  3. min 70%-75%
  4. min 75%-80%
  5. min 80%-85%
  10 min 85%-94%
  Interventions: Procedure: Titration of oxygen during newborn resuscitation in delivery room
- Traditional Oxygen strategy ( TOX) (Active Comparator): Resuscitation for TOX infants was started with 100% O2 and adjusted every 30 seconds by 10% to meet the target oxygen saturation range of 85-94%
  Interventions: Procedure: Titration of oxygen during newborn resuscitation in delivery room

INTERVENTIONS:
Procedure: Titration of oxygen during newborn resuscitation in delivery room

SUMMARY:
Preterm infants are born with immature lungs and often require help with breathing shortly after birth. This traditionally involves administering 100% oxygen. Unfortunately, delivery of high oxygen concentrations leads to the production of free radicals that can injure many organ systems. Term and near-term newborns deprived of oxygen during or prior to birth respond as well or better to resuscitation with room air (21% oxygen) compared to 100% oxygen. However, a static concentration of 21% oxygen may be inappropriate for preterm infants with lung disease.Purpose of the study is to investigate if preterm neonates where resuscitation is initiated with 21% fiO2 and adjusted to meet transitional goal saturations (Limited oxygen strategy or LOX) would have less oxidative stress as measured by the oxidative balance ratio of biological antioxidant potential/total hydroperoxide compared to infants where resuscitation is initiated with pure oxygen and titrated for targeted saturations of 85-94% (Traditional oxygen strategy or TOX). Secondary outcomes of interest included need for other delivery room resuscitation measures, respiratory support and ventilation/oxygenation status upon neonatal intensive care unit (NICU) admission, survival to hospital discharge, bronchopulmonary dysplasia and other short-term morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Inborn
* Gestation age 24 0/7 to 34 6/7
* Need for active resuscitation

Exclusion Criteria:

* Prenatally diagnosed cyanotic congenital heart disease
* Non-viable newborns
* Precipitous delivery and resuscitation team not present in the delivery room to initiate resuscitation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Reduction in mean oxidative balance ratio at 1 hour of life | Cord blood and at 1 hour of life
  Total hydroperoxide(TH), Biological antioxidant potential (BAP)were measured at 1 hour of life in all preterm infants. Oxidative balance ratio was calculated from this formula. Oxidative balance ratio = BAP/TH.

SECONDARY OUTCOMES:
Total oxygen load used during active resuscitation | First 10 minutes of life
Saturations achieved during first 10 minutes of life | First 10 minutes of life
Significant bradycardia ( HR<60 beats per minute) after 90 seconds in either group during active resuscitation | First 10 minutes of life
Time spent with saturation above 94% during active resuscitation | First 10 minutes of life
Need for respiratory support in the delivery room | First 10 minutes of life
Bronchopulmonary dysplasia | 36 weeks postconceptional age
Length of hospitalization | From date of randomization to date of discharge, expected average of 8 weeks
Retinopathy of Prematurity | 40 weeks postconceptional age
Neonatal mortality | 28 days of life
Death before discharge | From date of randomization to date of discharge, expected average of 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vishal S Kapadia, MD, Principal Investigator — UT Southwestern; Myra H Wyckoff, MD, Principal Investigator — UT Southwestern
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

REFERENCES:
- [Derived] Kapadia VS, Chalak LF, Sparks JE, Allen JR, Savani RC, Wyckoff MH. Resuscitation of preterm neonates with limited versus high oxygen strategy. Pediatrics. 2013 Dec;132(6):e1488-96. doi: 10.1542/peds.2013-0978. Epub 2013 Nov 11. PMID 24218465